CLINICAL TRIAL: NCT01543698
Title: A Phase Ib/II, Multicenter, Open-label, Dose Escalation Study of LGX818 in Combination With MEK162 in Adult Patients With BRAF V600 - Dependent Advanced Solid Tumors
Brief Title: A Phase Ib/II Study of LGX818 in Combination With MEK162 in Adult Patients With BRAF Dependent Advanced Solid Tumors
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CMEK162X2110; C4221005 (Other: Alias Study Number); 2011-005875-17 (EudraCT Number)
Record Dates: First submitted 2012-02-01; First posted 2012-03-05 (Estimated); Results first posted 2024-03-13 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-02

CONDITIONS: Solid Tumors Harboring a BRAF V600 Mutation
Keywords: Advanced solid tumor,; BRAF V600 mutation
MeSH Terms: interventions — encorafenib; binimetinib; ribociclib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- dual combination (Experimental): LGX818 QD and MEK162 BID
  Interventions: Drug: LGX818; Drug: MEK162
- triple combination (Experimental): LGX818 QD and MEK162 BID and LEE011 QD 3 weeks on, 1 week off.
  Interventions: Drug: LGX818; Drug: MEK162; Drug: LEE011

INTERVENTIONS:
Drug: LGX818
Drug: MEK162
Drug: LEE011
  Arms: triple combination

SUMMARY:
This is a multi-center, open-label, dose finding, Phase Ib dose escalation study to estimate the MTD(s) and/or RP2D(s) for the dual combination of LGX818 and MEK162 and the triple combination of LGX818 and MEK162 and LEE011, followed each independently by a Phase II part to assess the clinical efficacy and to further assess the safety of the combinations in selected patient populations. Oral LGX818 and MEK162 will be administered on a continuous schedule. Oral LEE011 will be administered once daily on a three weeks on, one week off schedule. Patients will be treated until progression of disease, unacceptable toxicity develops, or withdrawal of informed consent, whichever occurs first. A cycle is defined as 28 days. The dose escalation parts of the trial will be conducted in adult patients with BRAF V600-dependent advanced solid tumors and is expected to enroll at least 18 patients for the dual combination and at least 12 patients for the triple combination. The dose escalation will be guided by a Bayesian logistic regression model (BLRM). Following MTD/RP2D declaration, patients will be enrolled in three Phase II arms for the dual combination and one Phase II arm for the triple combination. All patients will be followed for 30 days for safety assessments after study drugs discontinuation. All patients enrolled in the Phase II part of the study will be followed for survival.

ELIGIBILITY:
Inclusion Criteria:

Histologically confirmed diagnosis of locally advanced or metastatic melanoma (stage IIIB to IV per American Joint Committee on Cancer [AJCC]), or confirmed diagnosis of non-resectable advanced metastatic colorectal cancer (mCRC), or any other indication upon agreement with the Sponsor, whose disease has progressed despite previous antineoplastic therapy or for whom no further effective standard therapy is available

* Written documentation of BRAF V600E mutation, or any other BRAF V600 mutation
* Evidence of measurable disease as determined by RECIST v1.1
* World Health Organization (WHO) Performance Status ≤ 2
* Negative serum pregnancy test within 72 hours prior to the first study dose in all women of childbearing potential

Exclusion Criteria:

Progressive disease following prior treatment with RAF-inhibitors in combination with MEK-inhibitors

* Symptomatic or untreated leptomeningeal disease
* Symptomatic brain metastases. Patients are not permitted to receive enzyme inducing anti-epileptic drugs
* Known acute or chronic pancreatitis
* History or current evidence of retinal disease, retinal vein occlusion or ophthalmopathy
* Clinically significant cardiac disease
* Patients with abnormal laboratory values at Screening/baseline
* Impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of oral LGX818/MEK162
* Previous or concurrent malignancy
* Pregnant or nursing (lactating) women
* For addition of LEE011 in the triple combination, congenital long QT syndrome or family history of unexpected sudden cardiac death and/or hypokalemia CTCAE Grade ≥ 3, brain metastases at baseline, abnormal coagulation results PT/INR >1.5 x ULN or aPTT >1.5 x ULN.

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 189 (Actual)
Dates: Start 2012-05-28 (Actual); Primary Completion 2023-03-09 (Actual); Study Completion 2023-03-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (26):
- United States (6):
  - H. Lee Moffitt Cancer Center & Research Institute, Inc., Tampa, Florida
  - Moffitt McKinley Outpatient Center, Tampa, Florida
  - Johns Hopkins Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Ophthalmic Consultants of Boston Inc (OCB), Boston, Massachusetts
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
- Australia (6):
  - Chris O'Brien Lifehouse Hospital, Camperdown, New South Wales
  - Melanoma Institute Australia, North Sydney, New South Wales
  - Westmead Hospital-Redbank Rd, Northmead, New South Wales
  - Westmead Hospital-Redbank Rd, Westmead, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Melanoma Institute Australia, North Sydney
- UZ Leuven- Gasthuisberg Campus, Leuven, Vlaams Brabant, Belgium
- Sir Mortimer B. Davis-Jewish General Hospital, Montreal, Quebec, Canada
- France (2):
  - Hôpital Saint louis, Paris
  - Service de radiologie - Hopital Saint Louis, Paris
- Italy (5):
  - IRCCS Fondazione Pascale, Naples, Campania
  - Azienda Ospedaliera Monaldi, Napoli, Campania
  - Azienda Ospedaliera Universitaria Federico II, Napoli, Campania
  - ASST Grande Ospedale Metropolitano Niguarda - Presidio Ospedaliero Ospedale Niguarda Ca' Granda, Milan
  - Istituto Nazionale per lo studio e la cura dei tumori Fondazione Giovanni Pascale, Napoli
- National Cancer Centre Singapore, Singapore, Singapore
- Spain (2):
  - Hospital Universitario Vall d'Hebrón - PPDS, Barcelona
  - Hospital Universitario HM Sanchinarro ? CIOCC, Madrid
- Switzerland (2):
  - University Hospital Zürich, Dermatology, Zurich-Airport, Canton of Zurich
  - Kantonsspital St. Gallen, Sankt Gallen

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Sullivan RJ, Weber J, Patel S, Dummer R, Carlino MS, Tan DSW, Lebbe C, Siena S, Elez E, Wollenberg L, Pickard MD, Sandor V, Ascierto PA. A Phase Ib/II Study of the BRAF Inhibitor Encorafenib Plus the MEK Inhibitor Binimetinib in Patients with BRAFV600E/K -mutant Solid Tumors. Clin Cancer Res. 2020 Oct 1;26(19):5102-5112. doi: 10.1158/1078-0432.CCR-19-3550. Epub 2020 Jul 15. PMID 32669376

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study had 2 Phases- 1b and 2. Phase 1b enrolled participants with V-raf murine sarcoma viral oncogene homolog B1 (BRAF) V600-dependent advanced solid tumors. Phase 2 enrolled participants with: BRAF V600 mutant metastatic colorectal cancer (mCRC) [Arm 1, dual]; BRAF V600 mutant melanoma who progressed after prior selective BRAF inhibitor treatment [Arm 2, dual]; metastatic BRAF mutant melanoma who were naïve to prior treatment with a selective BRAF inhibitor [Arm 3, dual]/ [Arm A, triple].
Pre-assignment Details: A total of 189 participants were enrolled. Phase 1 b: 47 participants for dual combination and 21 participants for triple combination. Phase 2: a) Dual combination- Arm 1 (mCRC) =11 participants; Arm 2 (prior BRAFi melanoma) =26 participants; Arm 3 (BRAFi-naïve melanoma) =42 participants and b) Triple combination- Arm A (BRAFi-naïve melanoma) =42 participants. Dual combination of LGX818 (encorafenib) and MEK162 (binimetinib) and triple combination of LGX818, MEK162 and LEE011 (ribociclib).
Groups:
- Phase 1b: Encorafenib 50 mg + Binimetinib 45 mg: Participants received Encorafenib 50 milligram (mg) once daily (QD) and Binimetinib 45 mg twice a daily (BID) orally 4 weeks till sponsor/investigator determined the maximum tolerated dose (MTD) and/or recommended phase II dose (RP2D), until disease progression, unacceptable toxicity or withdrawal of informed consent, whichever occurred first.
- Phase 1b: Encorafenib 100 mg+ Binimetinib 45 mg: Participants received Encorafenib 100 mg QD and Binimetinib 45 mg BID orally for 4 weeks till sponsor/investigator determined MTD and/or RP2D, until disease progression, unacceptable toxicity or withdrawal of informed consent, whichever occurred first.
- Phase 1b: Encorafenib 200 mg + Binimetinib 45 mg: Participants received Encorafenib 200 mg QD and Binimetinib 45 mg BID orally for 4 weeks till sponsor/investigator determined MTD and/or RP2D, until disease progression, unacceptable toxicity or withdrawal of informed consent, whichever occurred first.
- Phase 1b: Encorafenib 400 mg + Binimetinib 45 mg: Participants received Encorafenib 400 mg QD and Binimetinib 45 mg BID orally for 4 weeks till sponsor/investigator determined MTD and/or RP2D, until disease progression, unacceptable toxicity or withdrawal of informed consent, whichever occurred first.
- Phase 1b: Encorafenib 450 mg+ Binimetinib 45 mg: Participants received Encorafenib 450 mg QD and Binimetinib 45 mg BID orally for 4 weeks till sponsor/investigator determined MTD and/or RP2D, until disease progression, unacceptable toxicity or withdrawal of informed consent, whichever occurred first.
- Phase 1b: Encorafenib 600 mg + Binimetinib 45 mg: Participants received Encorafenib 600 mg QD and Binimetinib 45 mg BID orally for 4 weeks till sponsor/investigator determined MTD and/or RP2D, until disease progression, unacceptable toxicity or withdrawal of informed consent, whichever occurred first.
- Phase 1b: Encorafenib 800 mg + Binimetinib 45 mg: Participants received Encorafenib 800 mg QD and Binimetinib 45 mg BID orally for 4 weeks till sponsor/investigator determined MTD and/or RP2D, until disease progression, unacceptable toxicity or withdrawal of informed consent, whichever occurred first.
- Phase 1b: Encorafenib 200 mg+ Binimetinib 45 mg+ Ribociclib 100 mg: Participants received Encorafenib 200 mg QD and Binimetinib 45 mg BID orally on a continuous schedule of 4 weeks, and Ribociclib 100 mg BID orally for 3 weeks on, 1 week off schedule, till sponsor/investigator determined MTD and/or RP2D, until disease progression, unacceptable toxicity or withdrawal of informed consent, whichever occurred first.
- Phase 1b: Encorafenib 200 mg+ Binimetinib 45 mg+ Ribociclib 200 mg: Participants received Encorafenib 200 mg QD and Binimetinib 45 mg BID orally on a continuous schedule of 4 weeks, and Ribociclib 200 mg BID orally for 3 weeks on, 1 week off schedule, till sponsor/investigator determined MTD and/or RP2D, until disease progression, unacceptable toxicity or withdrawal of informed consent, whichever occurred first.
- Phase 1b: Encorafenib 200 mg+ Binimetinib 45 mg+ Ribociclib 400 mg: Participants received Encorafenib 200 mg QD and Binimetinib 45 mg BID orally on a continuous schedule of 4 weeks, and Ribociclib 400 mg BID orally for 3 weeks on, 1 week off schedule, till sponsor/investigator determined MTD and/or RP2D, until disease progression, unacceptable toxicity or withdrawal of informed consent, whichever occurred first.
- Phase 1b: Encorafenib 200 mg+ Binimetinib 45 mg + Ribociclib 600 mg: Participants received Encorafenib 200 mg QD and Binimetinib 45 mg BID orally on a continuous schedule of 4 weeks, and Ribociclib 600 mg BID orally for 3 weeks on, 1 week off schedule, till sponsor/investigator determined MTD and/or RP2D, until disease progression, unacceptable toxicity or withdrawal of informed consent, whichever occurred first.
- Phase 2: Arm 1 (mCRC): Encorafenib + Binimetinib; Phase 2: Arm 2 (Prior BRAFi Melanoma): Encorafenib + Binimetinib; Phase 2: Arm 3 (BRAFi-naïve Melanoma): Encorafenib + Binimetinib: Participants received Encorafenib at MTD (600 mg QD, permitted dose reduction to 450 mg QD) and Binimetinib 45 mg BID orally on a continuous schedule of 4 weeks until disease progression, unacceptable toxicity or withdrawal of informed consent, whichever occurred first.
- Phase 2: Arm A (BRAFi-naïve Melanoma): Encorafenib + Binimetinib + Ribociclib: Participants received Encorafenib 200 mg QD (MTD), Binimetinib 45 mg BID orally on a continuous schedule of 4 weeks, and Ribociclib 600 mg QD orally for 3 weeks on, 1 week off schedule until disease progression, unacceptable toxicity or withdrawal of informed consent, whichever occurred first.
Period: Phase 1b
Arm/Group | Phase 1b: Encorafenib 50 mg + Binimetinib 45 mg | Phase 1b: Encorafenib 100 mg+ Binimetinib 45 mg | Phase 1b: Encorafenib 200 mg + Binimetinib 45 mg | Phase 1b: Encorafenib 400 mg + Binimetinib 45 mg | Phase 1b: Encorafenib 450 mg+ Binimetinib 45 mg | Phase 1b: Encorafenib 600 mg + Binimetinib 45 mg | Phase 1b: Encorafenib 800 mg + Binimetinib 45 mg | Phase 1b: Encorafenib 200 mg+ Binimetinib 45 mg+ Ribociclib 100 mg | Phase 1b: Encorafenib 200 mg+ Binimetinib 45 mg+ Ribociclib 200 mg | Phase 1b: Encorafenib 200 mg+ Binimetinib 45 mg+ Ribociclib 400 mg | Phase 1b: Encorafenib 200 mg+ Binimetinib 45 mg + Ribociclib 600 mg | Phase 2: Arm 1 (mCRC): Encorafenib + Binimetinib | Phase 2: Arm 2 (Prior BRAFi Melanoma): Encorafenib + Binimetinib | Phase 2: Arm 3 (BRAFi-naïve Melanoma): Encorafenib + Binimetinib | Phase 2: Arm A (BRAFi-naïve Melanoma): Encorafenib + Binimetinib + Ribociclib
Started | 6 (Phase 1b participants received dual combination therapy.) | 5 (Phase 1b participants received dual combination therapy.) | 4 (Phase 1b participants received dual combination therapy.) | 5 (Phase 1b participants received dual combination therapy.) | 13 (Phase 1b participants received dual combination therapy.) | 8 (Phase 1b participants received dual combination therapy.) | 6 (Phase 1b participants received dual combination therapy.) | 4 (Phase 1b participants received triple combination therapy.) | 5 (Phase 1b participants received triple combination therapy.) | 6 (Phase 1b participants received triple combination therapy.) | 6 (Phase 1b participants received triple combination therapy.) | 0 (No participants in this arm enrolled in Phase 1b.) | 0 (No participants in this arm enrolled in Phase 1b.) | 0 (No participants in this arm enrolled in Phase 1b.) | 0 (No participants in this arm enrolled in Phase 1b.)
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 6 | 5 | 4 | 5 | 13 | 8 | 6 | 4 | 5 | 6 | 6 | 0 | 0 | 0 | 0
Not completed — Disease progression | 2 | 4 | 3 | 2 | 10 | 6 | 5 | 3 | 4 | 5 | 1 | 0 | 0 | 0 | 0
Not completed — Death | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 1 | 2 | 2 | 0 | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 0
Not completed — Administrative problems | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Phase 2
Arm/Group | Phase 1b: Encorafenib 50 mg + Binimetinib 45 mg | Phase 1b: Encorafenib 100 mg+ Binimetinib 45 mg | Phase 1b: Encorafenib 200 mg + Binimetinib 45 mg | Phase 1b: Encorafenib 400 mg + Binimetinib 45 mg | Phase 1b: Encorafenib 450 mg+ Binimetinib 45 mg | Phase 1b: Encorafenib 600 mg + Binimetinib 45 mg | Phase 1b: Encorafenib 800 mg + Binimetinib 45 mg | Phase 1b: Encorafenib 200 mg+ Binimetinib 45 mg+ Ribociclib 100 mg | Phase 1b: Encorafenib 200 mg+ Binimetinib 45 mg+ Ribociclib 200 mg | Phase 1b: Encorafenib 200 mg+ Binimetinib 45 mg+ Ribociclib 400 mg | Phase 1b: Encorafenib 200 mg+ Binimetinib 45 mg + Ribociclib 600 mg | Phase 2: Arm 1 (mCRC): Encorafenib + Binimetinib | Phase 2: Arm 2 (Prior BRAFi Melanoma): Encorafenib + Binimetinib | Phase 2: Arm 3 (BRAFi-naïve Melanoma): Encorafenib + Binimetinib | Phase 2: Arm A (BRAFi-naïve Melanoma): Encorafenib + Binimetinib + Ribociclib
Started | 0 (No participants in this arm enrolled in Phase 2.) | 0 (No participants in this arm enrolled in Phase 2.) | 0 (No participants in this arm enrolled in Phase 2.) | 0 (No participants in this arm enrolled in Phase 2.) | 0 (No participants in this arm enrolled in Phase 2.) | 0 (No participants in this arm enrolled in Phase 2.) | 0 (No participants in this arm enrolled in Phase 2.) | 0 (No participants in this arm enrolled in Phase 2.) | 0 (No participants in this arm enrolled in Phase 2.) | 0 (No participants in this arm enrolled in Phase 2.) | 0 (No participants in this arm enrolled in Phase 2.) | 11 (Phase 2 participants received dual combination therapy.) | 26 (Phase 2 participants received dual combination therapy.) | 42 (Phase 2 participants received dual combination therapy.) | 42 (Phase 2 participants received triple combination therapy.)
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 11 | 26 | 42 | 42
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Disease progression | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 10 | 21 | 30 | 25
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Not completed — Administrative problems | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 5 | 14

BASELINE CHARACTERISTICS:
Population: Safety set included all participants who received at least one dose of Encorafenib or Binimetinib or Ribociclib and had at least one valid post-baseline safety assessment.
Groups:
- Phase 1b: Encorafenib 50 mg + Binimetinib 45 mg: Participants received Encorafenib 50 mg QD and Binimetinib 45 mg BID orally on a schedule of continuous 4 weeks.
- Phase 1b: Encorafenib 100 mg+ Binimetinib 45 mg: Participants received Encorafenib 100 mg QD and Binimetinib 45 mg BID orally on a schedule of continuous 4 weeks.
- Phase 1b: Encorafenib 200 mg + Binimetinib 45 mg: Participants received Encorafenib 200 mg QD and Binimetinib 45 mg BID orally on a schedule of continuous 4 weeks.
- Phase 1b: Encorafenib 400 mg + Binimetinib 45 mg: Participants received Encorafenib 400 mg QD and Binimetinib 45 mg BID orally on a schedule of continuous 4 weeks.
- Phase 1b: Encorafenib 450 mg+ Binimetinib 45 mg: Participants received Encorafenib 450 mg QD and Binimetinib 45 mg BID orally on a schedule of continuous 4 weeks.
- Phase 1b: Encorafenib 600 mg + Binimetinib 45 mg: Participants received Encorafenib 600 mg QD and Binimetinib 45 mg BID orally on a schedule of continuous 4 weeks.
- Phase 1b: Encorafenib 800 mg + Binimetinib 45 mg: Participants received Encorafenib 800 mg QD and Binimetinib 45 mg BID orally on a schedule of continuous 4 weeks.
- Phase 1b: Encorafenib 200 mg+ Binimetinib 45 mg+ Ribociclib 100 mg: Participants received Encorafenib 200 mg QD, Binimetinib 45 mg BID orally on a schedule of continuous 4 weeks and Ribociclib 100 mg QD orally for 3 weeks on, 1 week off schedule.
- Phase 1b: Encorafenib 200 mg+ Binimetinib 45 mg+ Ribociclib 200 mg: Participants received Encorafenib 200 mg QD, Binimetinib 45 mg BID orally on a schedule of continuous 4 weeks and Ribociclib 200 mg QD orally for 3 weeks on, 1 week off schedule.
- Phase 1b: Encorafenib 200 mg+ Binimetinib 45 mg+ Ribociclib 400 mg: Participants received Encorafenib 200 mg QD, Binimetinib 45 mg BID orally on a schedule of continuous 4 weeks and Ribociclib 400 mg QD orally for 3 weeks on, 1 week off schedule.
- Phase 1b: Encorafenib 200 mg+ Binimetinib 45 mg + Ribociclib 600 mg: Participants received Encorafenib 200 mg QD, Binimetinib 45 mg BID orally on a schedule of continuous 4 weeks and Ribociclib 600 mg QD orally for 3 weeks on, 1 week off schedule.
- Phase 2: Arm 2 (Prior BRAFi Melanoma): Encorafenib + Binimetinib; Phase 2: Arm 3 (BRAFi-naïve Melanoma): Encorafenib + Binimetinib: Participants received Encorafenib at MTD (600 mg QD, permitted dose reduction to 450 mg QD) and Binimetinib 45 mg BID orally on a continuous schedule of 4 weeks.
- Phase 2: Arm A (BRAFi-naïve Melanoma): Encorafenib + Binimetinib + Ribociclib: Participants received Encorafenib 200 mg QD (MTD), Binimetinib 45 mg BID orally on a continuous schedule of 4 weeks, and Ribociclib 600 mg QD orally for 3 weeks on, 1 week off schedule.
- Total: Total of all reporting groups
Arm/Group | Phase 1b: Encorafenib 50 mg + Binimetinib 45 mg | Phase 1b: Encorafenib 100 mg+ Binimetinib 45 mg | Phase 1b: Encorafenib 200 mg + Binimetinib 45 mg | Phase 1b: Encorafenib 400 mg + Binimetinib 45 mg | Phase 1b: Encorafenib 450 mg+ Binimetinib 45 mg | Phase 1b: Encorafenib 600 mg + Binimetinib 45 mg | Phase 1b: Encorafenib 800 mg + Binimetinib 45 mg | Phase 1b: Encorafenib 200 mg+ Binimetinib 45 mg+ Ribociclib 100 mg | Phase 1b: Encorafenib 200 mg+ Binimetinib 45 mg+ Ribociclib 200 mg | Phase 1b: Encorafenib 200 mg+ Binimetinib 45 mg+ Ribociclib 400 mg | Phase 1b: Encorafenib 200 mg+ Binimetinib 45 mg + Ribociclib 600 mg | Phase 2: Arm 1 (mCRC): Encorafenib + Binimetinib | Phase 2: Arm 2 (Prior BRAFi Melanoma): Encorafenib + Binimetinib | Phase 2: Arm 3 (BRAFi-naïve Melanoma): Encorafenib + Binimetinib | Phase 2: Arm A (BRAFi-naïve Melanoma): Encorafenib + Binimetinib + Ribociclib | Total
Number analyzed (Participants) | 6 | 5 | 4 | 5 | 13 | 8 | 6 | 4 | 5 | 6 | 6 | 11 | 26 | 42 | 42 | 189
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 4 | 4 | 4 | 10 | 6 | 5 | 4 | 4 | 3 | 6 | 9 | 22 | 33 | 32 | 149
  >=65 years | 3 | 1 | 0 | 1 | 3 | 2 | 1 | 0 | 1 | 3 | 0 | 2 | 4 | 9 | 10 | 40
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 4 | 1 | 5 | 3 | 4 | 1 | 4 | 1 | 4 | 3 | 11 | 12 | 19 | 77
  Male | 4 | 2 | 0 | 4 | 8 | 5 | 2 | 3 | 1 | 5 | 2 | 8 | 15 | 30 | 23 | 112
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Caucasian | 4 | 5 | 2 | 5 | 12 | 8 | 6 | 4 | 5 | 6 | 6 | 11 | 24 | 37 | 42 | 177
  Race: Asian | 2 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 6
  Race: Other | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 5 | 0 | 6
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Hispanic/Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 4
  Ethnicity: Chinese | 2 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5
  Ethnicity: Other | 4 | 5 | 2 | 5 | 12 | 8 | 6 | 4 | 5 | 6 | 6 | 11 | 24 | 41 | 41 | 180

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose Limiting Toxicities (DLTs): Phase 1b
Description: DLT was defined as an adverse event or abnormal laboratory value assessed as at least possibly related to the study medication, as clinically relevant, as unrelated to disease, disease progression, inter-current illness, or concomitant medications, which occurred (less than equal to) <=28 days following the first dose of LGX818 and MEK162 or LGX818 and MEK162 and LEE011 (cycle 1) and met the defined criteria for the study.
Time Frame: Phase 1b: Cycle 1 (28 days following the first dose of LGX818 and MEK162 or LGX818 and MEK162 and LEE011)
Population: Dose Determining Set (DDS) included all Phase 1b participants from the safety set who either completed a minimum exposure requirement and had sufficient safety evaluations or discontinued prematurely due to a DLT. All participants reported under "Number of Participants Analyzed" contributed data to this outcome measure.
Measure: Count of Participants; unit: Participants
Groups:
- Phase 1b: Encorafenib 100 mg + Binimetinib 45 mg: Participants received Encorafenib 100 mg QD and Binimetinib 45 mg BID orally on a schedule of continuous 4 weeks.
- Phase 1b: Encorafenib 450 mg + Binimetinib 45 mg: Participants received Encorafenib 450 mg QD and Binimetinib 45 mg BID orally on a schedule of continuous 4 weeks.
- Phase 1b: Encorafenib 200 mg + Binimetinib 45 mg+ Ribociclib 100 mg: Participants received Encorafenib 200 mg QD, Binimetinib 45 mg BID orally on a schedule of continuous 4 weeks and Ribociclib 100 mg QD orally for 3 weeks on,1 week off schedule.
- Phase 1b: Encorafenib 200 mg + Binimetinib 45 mg + Ribociclib 200 mg: Participants received Encorafenib 200 mg QD, Binimetinib 45 mg BID orally on a schedule of continuous 4 weeks and Ribociclib 200 mg QD orally for 3 weeks on,1 week off schedule.
- Phase 1b: Encorafenib 200 mg+ Binimetinib 45 mg+ Ribociclib 400 mg: Participants received Encorafenib 200 mg QD, Binimetinib 45 mg BID orally on a schedule of continuous 4 weeks and Ribociclib 400 mg QD orally for 3 weeks on,1 week off schedule.
- Phase 1b: Encorafenib 200 mg + Binimetinib 45 mg+ Ribociclib 600 mg: Participants received Encorafenib 200 mg QD, Binimetinib 45 mg BID orally on a schedule of continuous 4 weeks and Ribociclib 600 mg QD orally for 3 weeks on,1 week off schedule.
Arm/Group | Phase 1b: Encorafenib 50 mg + Binimetinib 45 mg | Phase 1b: Encorafenib 100 mg + Binimetinib 45 mg | Phase 1b: Encorafenib 200 mg + Binimetinib 45 mg | Phase 1b: Encorafenib 400 mg + Binimetinib 45 mg | Phase 1b: Encorafenib 450 mg + Binimetinib 45 mg | Phase 1b: Encorafenib 600 mg + Binimetinib 45 mg | Phase 1b: Encorafenib 800 mg + Binimetinib 45 mg | Phase 1b: Encorafenib 200 mg + Binimetinib 45 mg+ Ribociclib 100 mg | Phase 1b: Encorafenib 200 mg + Binimetinib 45 mg + Ribociclib 200 mg | Phase 1b: Encorafenib 200 mg+ Binimetinib 45 mg+ Ribociclib 400 mg | Phase 1b: Encorafenib 200 mg + Binimetinib 45 mg+ Ribociclib 600 mg
Number analyzed (Participants) | 6 | 5 | 2 | 4 | 13 | 8 | 6 | 4 | 5 | 5 | 5
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0

2. Primary Outcome: Disease Control Rate (DCR) at Week 16: Phase 2, Arm 1 (mCRC Participants)
Description: DCR was defined as percentage of participants with a best overall response of complete response (CR), partial response (PR) or stable disease (SD). As per Response Evaluation Criteria in Solid tumors Response Evaluation Criteria in Solid Tumors (RECIST) v1.1: CR was defined as complete disappearance of all target lesions and non-target disease. All nodes, both target and non-target, must have a reduction in short axis less than (<)10 millimeter [mm]). PR was defined as more than equal to (>=) 30 percent (%) decrease under baseline of sum of diameters of all target lesions taking as reference the baseline sum of diameters. SD was defined as neither sufficient shrinkage to qualify for PR or CR nor an increase in lesions which would qualify for progressive disease (PD).
Time Frame: Phase 2: Week 16
Population: Full Analysis Set (FAS) included all participants who received at least one dose of LGX818 or MEK162 or LEE011.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Phase 2: Arm 1 (mCRC): Encorafenib + Binimetinib
Number analyzed (Participants) | 11
Percentage of participants | 63.6 [30.8 to 89.1]

3. Primary Outcome: Objective Response Rate (ORR): Phase 2, Arms 2, 3 and A
Description: ORR was defined as the percentage of participants with a best overall response of CR or PR. As per RECIST v1.1, CR was defined as complete disappearance of all target lesions and non-target disease. All nodes, both target and non-target, must have a reduction in short axis <10 mm. PR was defined as >= 30% decrease under baseline of sum of diameters of all target lesions taking as reference the baseline sum of diameters.
Time Frame: Phase 2: From Day 1 of dosing till complete response or partial response achieved (maximum exposure of treatment for Phase 2 was 111.5 months]
Population: FAS included all participants who received at least one dose of LGX818 or MEK162 or LEE011.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Phase 2: Arm 2 (Prior BRAFi Melanoma): Encorafenib + Binimetinib | Phase 2: Arm 3 (BRAFi-naïve Melanoma): Encorafenib + Binimetinib | Phase 2: Arm A (BRAFi-naïve Melanoma): Encorafenib + Binimetinib + Ribociclib
Number analyzed (Participants) | 26 | 42 | 42
Percentage of participants | 42.3 [23.4 to 63.1] | 66.7 [50.5 to 80.4] | 59.5 [43.3 to 74.4]

4. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs): Overall Grades and AEs of Grade 3/4: Phase 1b
Description: An AE was any untoward medical occurrence in a participant or clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. TEAEs were those events with onset dates occurring during the on-treatment period (the time from the Day 1 up to 30 days after last dose). AEs were graded according to National Cancer Institute's Common Terminology Criteria for Adverse Events (CTCAE) version 4.03 as Grade 1 indicates Mild AE, Grade 2 indicates Moderate AE, Grade 3 indicates severe AE, and grade 4 indicates life-threatening consequences; urgent intervention indicated. Grade 5 indicates death related to AE.
Time Frame: Phase 1b: Day 1 up to 30 days after last dose (maximum treatment exposure for Phase 1b was 118.3 months)
Population: Safety set included all participants who received at least one dose of LGX818 or MEK162 or LEE011 and had at least one valid post-baseline safety assessment.
Measure: Count of Participants; unit: Participants
Groups:
- Phase 1b: Encorafenib 800 mg+ Binimetinib 45 mg: Participants received Encorafenib 800 mg QD and Binimetinib 45 mg BID orally on a schedule of continuous 4 weeks.
- Phase 1b: Encorafenib 200 mg+ Binimetinib 45 mg+ Ribociclib 200 mg: Participants received Encorafenib 200 mg QD, Binimetinib 45 mg BID orally on a schedule of continuous 4 weeks and Ribociclib 200 mg QD orally for 3 weeks on,1 week off schedule.
- Phase 1b: Encorafenib 200 mg + Binimetinib 45 mg+ Ribociclib 400 mg: Participants received Encorafenib 200 mg QD, Binimetinib 45 mg BID orally on a schedule of continuous 4 weeks and Ribociclib 400 mg QD orally for 3 weeks on,1 week off schedule.
- Phase 1b: Encorafenib 200 mg+ Binimetinib 45 mg + Ribociclib 600 mg: Participants received Encorafenib 200 mg QD, Binimetinib 45 mg BID orally on a schedule of continuous 4 weeks and Ribociclib 600 mg QD orally for 3 weeks on,1 week off schedule.
Arm/Group | Phase 1b: Encorafenib 50 mg + Binimetinib 45 mg | Phase 1b: Encorafenib 100 mg+ Binimetinib 45 mg | Phase 1b: Encorafenib 200 mg + Binimetinib 45 mg | Phase 1b: Encorafenib 400 mg + Binimetinib 45 mg | Phase 1b: Encorafenib 450 mg + Binimetinib 45 mg | Phase 1b: Encorafenib 600 mg + Binimetinib 45 mg | Phase 1b: Encorafenib 800 mg+ Binimetinib 45 mg | Phase 1b: Encorafenib 200 mg + Binimetinib 45 mg+ Ribociclib 100 mg | Phase 1b: Encorafenib 200 mg+ Binimetinib 45 mg+ Ribociclib 200 mg | Phase 1b: Encorafenib 200 mg + Binimetinib 45 mg+ Ribociclib 400 mg | Phase 1b: Encorafenib 200 mg+ Binimetinib 45 mg + Ribociclib 600 mg
Number analyzed (Participants) | 6 | 5 | 4 | 5 | 13 | 8 | 6 | 4 | 5 | 6 | 6
Participants
  Overall Grades | 6 | 5 | 4 | 5 | 13 | 8 | 6 | 4 | 5 | 6 | 6
  Grade 3/4 | 5 | 2 | 2 | 4 | 8 | 6 | 6 | 4 | 4 | 6 | 6

5. Secondary Outcome: Number of Participants With TEAEs: Overall Grades and AEs of Grade 3/4: Phase 2
Description: An AE was any untoward medical occurrence in a participant or clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. TEAEs were those events with onset dates occurring during the on-treatment period (the time from the Day 1 up to 30 days after last dose). AEs were graded according to CTCAE version 4.03 as Grade 1 indicates Mild AE, Grade 2 indicates Moderate AE, Grade 3 indicates severe AE, and grade 4 indicates life-threatening consequences; urgent intervention indicated. Grade 5 indicates death related to AE.
Time Frame: Phase 2: Day 1 up to 30 days after last dose (maximum treatment exposure for Phase 2 was 111.5 months)
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2: Arm 1 (mCRC): Encorafenib + Binimetinib | Phase 2: Arm 2 (Prior BRAFi Melanoma): Encorafenib + Binimetinib | Phase 2: Arm 3 (BRAFi-naïve Melanoma): Encorafenib + Binimetinib | Phase 2: Arm A (BRAFi-naïve Melanoma): Encorafenib + Binimetinib + Ribociclib
Number analyzed (Participants) | 11 | 26 | 42 | 42
Participants
  Overall Grades | 11 | 26 | 42 | 42
  Grade 3/4 | 5 | 15 | 27 | 34

6. Secondary Outcome: Area Under the Concentration-time Curve From Time Zero to Infinity With Extrapolation of the Terminal Phase (AUCinf) of Encorafenib, Binimetinib, Ribociclib, Metabolite of Binimetinib and Ribociclib: Phase 1b
Description: AUCinf was reported in unit of measure as hour*nanogram per millilitre (h*ng/mL).
Time Frame: Phase 1b: Pre dose, 0.5,1.5,2.5,4,6,8 and 24 hours (hr) post dose on Day 1 of Cycle 1
Population: FAS evaluated. All participants reported under "Number of Participants Analyzed" contributed data to the table; however, may not have evaluable data for every row. Here, "Number Analyzed" signifies number of participants evaluable for specified rows.
Measure: Mean (Standard Deviation); unit: h*ng/mL
Groups:
- Phase 1b: Encorafenib 50 mg+ Binimetinib 45 mg: Participants received Encorafenib 50 mg QD and Binimetinib 45 mg BID orally on a schedule of continuous 4 weeks.
- Phase 1b: Encorafenib 200 mg+ Binimetinib 45 mg: Participants received Encorafenib 200 mg QD and Binimetinib 45 mg BID orally on a schedule of continuous 4 weeks.
- Phase 1b: Encorafenib 400 mg+ Binimetinib 45 mg: Participants received Encorafenib 400 mg QD and Binimetinib 45 mg BID orally on a schedule of continuous 4 weeks.
- Phase 1b: Encorafenib 200 mg+ Binimetinib 45 mg + Ribociclib 100 mg: Participants received Encorafenib 200 mg QD, Binimetinib 45 mg BID orally on a schedule of continuous 4 weeks and Ribociclib 100 mg QD orally for 3 weeks on,1 week off schedule.
- Phase 1b: Encorafenib 200 mg + Binimetinib 45 mg+ Ribociclib 200 mg: Participants received Encorafenib 200 mg QD, Binimetinib 45 mg BID orally on a schedule of continuous 4 weeks and Ribociclib 200 mg QD orally for 3 weeks on,1 week off schedule.
- Phase 1b: Encorafenib 200 mg+ Binimetinib 45 mg+ Ribociclib 600 mg: Participants received Encorafenib 200 mg QD, Binimetinib 45 mg BID orally on a schedule of continuous 4 weeks and Ribociclib 600 mg QD orally for 3 weeks on,1 week off schedule.
Arm/Group | Phase 1b: Encorafenib 50 mg+ Binimetinib 45 mg | Phase 1b: Encorafenib 100 mg+ Binimetinib 45 mg | Phase 1b: Encorafenib 200 mg+ Binimetinib 45 mg | Phase 1b: Encorafenib 400 mg+ Binimetinib 45 mg | Phase 1b: Encorafenib 450 mg + Binimetinib 45 mg | Phase 1b: Encorafenib 600 mg + Binimetinib 45 mg | Phase 1b: Encorafenib 800 mg+ Binimetinib 45 mg | Phase 1b: Encorafenib 200 mg+ Binimetinib 45 mg + Ribociclib 100 mg | Phase 1b: Encorafenib 200 mg + Binimetinib 45 mg+ Ribociclib 200 mg | Phase 1b: Encorafenib 200 mg+ Binimetinib 45 mg+ Ribociclib 400 mg | Phase 1b: Encorafenib 200 mg+ Binimetinib 45 mg+ Ribociclib 600 mg
Number analyzed (Participants) | 6 | 5 | 4 | 5 | 13 | 8 | 6 | 4 | 5 | 6 | 6
h*ng/mL
  Encorafenib: number analyzed (Participants) | 6 | 5 | 4 | 4 | 13 | 7 | 5 | 4 | 4 | 3 | 5
  Encorafenib | 3740 (2350) | 11700 (6200) | 22000 (9790) | 42000 (23600) | 36700 (19400) | 57400 (27100) | 40200 (12100) | 15000 (7360) | 9960 (5940) | 18900 (9900) | 17400 (9480)
  Binimetinib: number analyzed (Participants) | 5 | 4 | 3 | 3 | 11 | 7 | 4 | 4 | 4 | 3 | 4
  Binimetinib | 2190 (1350) | 1930 (529) | 3730 (2250) | 1960 (1140) | 2750 (1490) | 3090 (1600) | 2340 (462) | 2160 (1580) | 3000 (932) | 3110 (1450) | 2970 (458)
  Ribociclib: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 5 | 4 | 4
  Ribociclib |  |  |  |  |  |  |  | 1040 (665) | 3030 (1600) | 7930 (5180) | 18200 (10400)
  Metabolite of Binimetinib: number analyzed (Participants) | 5 | 3 | 2 | 3 | 9 | 5 | 4 | 3 | 4 | 0 | 4
  Metabolite of Binimetinib | 321 (225) | 271 (28.9) | 631 (296) | 275 (121) | 361 (184) | 449 (302) | 361 (78.1) | 173 (55.6) | 337 (29.2) |  | 239 (79.1)
  Metabolite of Ribociclib: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 1 | 1
  Metabolite of Ribociclib |  |  |  |  |  |  |  | 194 (NA) — Standard deviation could not be calculated as only 1 participant was evaluable. | 601 (225) | 1340 (NA) — Standard deviation could not be calculated as only 1 participant was evaluable. | 2160 (NA) — Standard deviation could not be calculated as only 1 participant was evaluable.

7. Secondary Outcome: Area Under the Concentration-Time Curve From Time Zero to the Last Measurable Concentration Sampling Time (AUClast) of Encorafenib, Binimetinib, Ribociclib, Metabolite of Binimetinib and Ribociclib: Phase 1b
Time Frame: Phase 1b: Pre dose, 0.5,1.5,2.5,4,6,8 and 24 hr post dose on Day 1 of Cycle 1
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: h*ng/mL
Groups:
- Phase 1b: Encorafenib 600 mg+ Binimetinib 45 mg: Participants received Encorafenib 600 mg QD and Binimetinib 45 mg BID orally on a schedule of continuous 4 weeks.
- Phase 1b: Encorafenib 200 mg+ Binimetinib 45 mg+ Ribociclib 100 mg: Participants received Encorafenib 200 mg QD, Binimetinib 45 mg BID orally on a schedule of continuous 4 weeks and Ribociclib 100 mg QD orally for 3 weeks on,1 week off schedule.
Arm/Group | Phase 1b: Encorafenib 50 mg+ Binimetinib 45 mg | Phase 1b: Encorafenib 100 mg+ Binimetinib 45 mg | Phase 1b: Encorafenib 200 mg+ Binimetinib 45 mg | Phase 1b: Encorafenib 400 mg+ Binimetinib 45 mg | Phase 1b: Encorafenib 450 mg + Binimetinib 45 mg | Phase 1b: Encorafenib 600 mg+ Binimetinib 45 mg | Phase 1b: Encorafenib 800 mg+ Binimetinib 45 mg | Phase 1b: Encorafenib 200 mg+ Binimetinib 45 mg+ Ribociclib 100 mg | Phase 1b: Encorafenib 200 mg + Binimetinib 45 mg+ Ribociclib 200 mg | Phase 1b: Encorafenib 200 mg+ Binimetinib 45 mg+ Ribociclib 400 mg | Phase 1b: Encorafenib 200 mg+ Binimetinib 45 mg+ Ribociclib 600 mg
Number analyzed (Participants) | 6 | 5 | 4 | 5 | 13 | 8 | 6 | 4 | 5 | 6 | 6
h*ng/mL
  Encorafenib: number analyzed (Participants) | 6 | 5 | 4 | 4 | 13 | 7 | 6 | 4 | 5 | 6 | 6
  Encorafenib | 3690 (2340) | 11500 (6070) | 22000 (9750) | 40200 (21700) | 36100 (19300) | 57000 (26800) | 38100 (11800) | 11400 (4530) | 9280 (4190) | 12700 (5020) | 15800 (7160)
  Binimetinib: number analyzed (Participants) | 6 | 5 | 3 | 4 | 13 | 7 | 4 | 4 | 5 | 6 | 6
  Binimetinib | 1990 (1130) | 1990 (715) | 3300 (1990) | 1870 (867) | 2330 (1220) | 2790 (1480) | 2120 (478) | 1520 (663) | 2470 (878) | 2020 (843) | 2320 (635)
  Ribociclib: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 5 | 6 | 6
  Ribociclib |  |  |  |  |  |  |  | 806 (549) | 2550 (1280) | 6700 (3720) | 14500 (7490)
  Metabolite of Binimetinib: number analyzed (Participants) | 6 | 5 | 3 | 4 | 13 | 7 | 4 | 4 | 5 | 6 | 6
  Metabolite of Binimetinib | 276 (184) | 280 (50.5) | 372 (320) | 241 (82.5) | 287 (122) | 340 (244) | 307 (78.4) | 156 (53.8) | 259 (54.3) | 168 (109) | 161 (81.9)
  Metabolite of Ribociclib: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 5 | 6 | 6
  Metabolite of Ribociclib |  |  |  |  |  |  |  | 81.4 (41.0) | 397 (145) | 758 (231) | 1200 (320)

8. Secondary Outcome: AUClast at Steady State (AUClast,ss) of Encorafenib, Binimetinib, Ribociclib, Metabolite of Binimetinib and Ribociclib: Phase 1b
Time Frame: Phase 1b: Pre dose,0.5,1.5, 2.5,4,6,8 and 24 hr post dose on Day 15 of Cycle 1
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Phase 1b: Encorafenib 50 mg+ Binimetinib 45 mg | Phase 1b: Encorafenib 100 mg+ Binimetinib 45 mg | Phase 1b: Encorafenib 200 mg+ Binimetinib 45 mg | Phase 1b: Encorafenib 400 mg+ Binimetinib 45 mg | Phase 1b: Encorafenib 450 mg+ Binimetinib 45 mg | Phase 1b: Encorafenib 600 mg+ Binimetinib 45 mg | Phase 1b: Encorafenib 800 mg+ Binimetinib 45 mg | Phase 1b: Encorafenib 200 mg+ Binimetinib 45 mg+ Ribociclib 100 mg | Phase 1b: Encorafenib 200 mg+ Binimetinib 45 mg+ Ribociclib 200 mg | Phase 1b: Encorafenib 200 mg+ Binimetinib 45 mg+ Ribociclib 400 mg | Phase 1b: Encorafenib 200 mg+ Binimetinib 45 mg+ Ribociclib 600 mg
Number analyzed (Participants) | 6 | 5 | 4 | 5 | 13 | 8 | 6 | 4 | 5 | 6 | 6
h*ng/mL
  Encorafenib: number analyzed (Participants) | 6 | 5 | 2 | 3 | 11 | 6 | 6 | 4 | 5 | 5 | 5
  Encorafenib | 2620 (1260) | 5510 (1280) | 4620 (1640) | 10200 (2280) | 15900 (8730) | 27300 (17900) | 25300 (7240) | 6310 (2340) | 8210 (2550) | 11800 (7000) | 15700 (6060)
  Binimetinib: number analyzed (Participants) | 6 | 5 | 2 | 4 | 11 | 6 | 5 | 4 | 4 | 5 | 5
  Binimetinib | 2950 (1380) | 2610 (873) | 2660 (1900) | 2110 (1220) | 2550 (901) | 2590 (1640) | 2540 (529) | 2180 (1180) | 2820 (954) | 2740 (1230) | 2970 (1180)
  Ribociclib: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 5 | 5 | 5
  Ribociclib |  |  |  |  |  |  |  | 462 (129) | 1520 (979) | 5620 (3730) | 10100 (2970)
  Metabolite of Binimetinib: number analyzed (Participants) | 6 | 5 | 2 | 4 | 11 | 6 | 5 | 4 | 4 | 5 | 5
  Metabolite of Binimetinib | 147 (152) | 173 (125) | 118 (70.7) | 119 (96.5) | 157 (104) | 132 (142) | 190 (79.8) | 149 (136) | 210 (68.4) | 176 (92.5) | 169 (48.5)
  Metabolite of Ribociclib: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 5 | 5 | 5
  Metabolite of Ribociclib |  |  |  |  |  |  |  | 255 (131) | 729 (267) | 2150 (399) | 3260 (891)

9. Secondary Outcome: Area Under the Concentration-Time Curve From Time Zero to Tau After First Dose (AUCtau) of Encorafenib, Binimetinib, Ribociclib, Metabolite of Binimetinib and Ribociclib: Phase 1b
Time Frame: Phase 1b: Pre dose, 0.5,1.5,2.5,4,6,8 and 24 hr post dose on Day 1 of Cycle 1
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: h*ng/mL
Groups:
- Phase 1b: Encorafenib 200 mg+ Binimetinib 45 mg + Ribociclib 400 mg: Participants received Encorafenib 200 mg QD, Binimetinib 45 mg BID orally on a schedule of continuous 4 weeks and Ribociclib 400 mg QD orally for 3 weeks on,1 week off schedule.
Arm/Group | Phase 1b: Encorafenib 50 mg+ Binimetinib 45 mg | Phase 1b: Encorafenib 100 mg + Binimetinib 45 mg | Phase 1b: Encorafenib 200 mg+ Binimetinib 45 mg | Phase 1b: Encorafenib 400 mg+ Binimetinib 45 mg | Phase 1b: Encorafenib 450 mg+ Binimetinib 45 mg | Phase 1b: Encorafenib 600 mg+ Binimetinib 45 mg | Phase 1b: Encorafenib 800 mg+ Binimetinib 45 mg | Phase 1b: Encorafenib 200 mg+ Binimetinib 45 mg+ Ribociclib 100 mg | Phase 1b: Encorafenib 200 mg+ Binimetinib 45 mg+ Ribociclib 200 mg | Phase 1b: Encorafenib 200 mg+ Binimetinib 45 mg + Ribociclib 400 mg | Phase 1b: Encorafenib 200 mg+ Binimetinib 45 mg+ Ribociclib 600 mg
Number analyzed (Participants) | 6 | 5 | 4 | 5 | 13 | 8 | 6 | 4 | 5 | 6 | 6
h*ng/mL
  Encorafenib: number analyzed (Participants) | 6 | 5 | 4 | 4 | 13 | 7 | 5 | 4 | 4 | 3 | 5
  Encorafenib | 3700 (2320) | 11500 (6070) | 22000 (9750) | 40200 (21700) | 36300 (19000) | 57000 (26800) | 40000 (12100) | 14800 (7140) | 9940 (5900) | 18700 (9730) | 17300 (9300)
  Binimetinib: number analyzed (Participants) | 5 | 4 | 3 | 3 | 11 | 7 | 4 | 4 | 4 | 3 | 4
  Binimetinib | 2130 (1330) | 1860 (532) | 3600 (2160) | 1890 (1110) | 2650 (1410) | 3010 (1560) | 2280 (477) | 1790 (979) | 2900 (939) | 2860 (1320) | 2900 (453)
  Ribociclib: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 5 | 6 | 6
  Ribociclib |  |  |  |  |  |  |  | 845 (504) | 2550 (1280) | 6700 (3720) | 14500 (7490)
  Metabolite of Binimetinib: number analyzed (Participants) | 5 | 3 | 2 | 3 | 9 | 5 | 4 | 3 | 4 | 0 | 4
  Metabolite of Binimetinib | 307 (222) | 265 (27.9) | 585 (304) | 257 (109) | 338 (162) | 430 (291) | 344 (82.0) | 152 (32.3) | 322 (23.5) |  | 230 (79.1)
  Metabolite of Ribociclib: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 5 | 6 | 6
  Metabolite of Ribociclib |  |  |  |  |  |  |  | 98.9 (25.9) | 397 (145) | 758 (231) | 1200 (320)

10. Secondary Outcome: AUCtau at Steady State (AUCtau,ss) of Encorafenib, Binimetinib and Ribociclib, Metabolite of Binimetinib and Ribociclib: Phase 1b
Time Frame: Phase 1b: Pre dose,0.5,1.5, 2.5,4,6,8 and 24 hr post dose on Day 15 of Cycle 1
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Phase 1b: Encorafenib 50 mg+ Binimetinib 45 mg | Phase 1b: Encorafenib 100 mg+ Binimetinib 45 mg | Phase 1b: Encorafenib 200 mg + Binimetinib 45 mg | Phase 1b: Encorafenib 400 mg+ Binimetinib 45 mg | Phase 1b: Encorafenib 450 mg + Binimetinib 45 mg | Phase 1b: Encorafenib 600 mg+ Binimetinib 45 mg | Phase 1b: Encorafenib 800 mg+ Binimetinib 45 mg | Phase 1b: Encorafenib 200 mg+ Binimetinib 45 mg+ Ribociclib 100 mg | Phase 1b: Encorafenib 200 mg + Binimetinib 45 mg+ Ribociclib 200 mg | Phase 1b: Encorafenib 200 mg+ Binimetinib 45 mg+ Ribociclib 400 mg | Phase 1b: Encorafenib 200 mg+ Binimetinib 45 mg + Ribociclib 600 mg
Number analyzed (Participants) | 6 | 5 | 4 | 5 | 13 | 8 | 6 | 4 | 5 | 6 | 6
h*ng/mL
  Encorafenib: number analyzed (Participants) | 6 | 5 | 2 | 3 | 11 | 6 | 6 | 4 | 5 | 5 | 5
  Encorafenib | 2620 (1260) | 5510 (1280) | 4620 (1640) | 10200 (2280) | 15900 (8730) | 27300 (17900) | 25300 (7240) | 6310 (2340) | 8210 (2550) | 11800 (7000) | 15700 (6060)
  Binimetinib: number analyzed (Participants) | 6 | 5 | 2 | 4 | 11 | 6 | 5 | 4 | 4 | 5 | 5
  Binimetinib | 2950 (1380) | 2610 (873) | 2660 (1900) | 2110 (1220) | 2550 (901) | 2590 (1640) | 2540 (529) | 2180 (1180) | 2820 (954) | 2740 (1230) | 2970 (1180)
  Ribociclib: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 5 | 5 | 5
  Ribociclib |  |  |  |  |  |  |  | 462 (129) | 1520 (979) | 5620 (3730) | 10100 (2970)
  Metabolite of Binimetinib: number analyzed (Participants) | 3 | 3 | 2 | 2 | 7 | 2 | 4 | 2 | 4 | 4 | 5
  Metabolite of Binimetinib | 261 (136) | 237 (107) | 126 (59.5) | 194 (75.8) | 221 (83.5) | 304 (77.7) | 225 (25.1) | 265 (33.4) | 219 (71.5) | 207 (69.7) | 175 (52.8)
  Metabolite of Ribociclib: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 5 | 5 | 5
  Metabolite of Ribociclib |  |  |  |  |  |  |  | 255 (131) | 729 (267) | 2150 (399) | 3260 (891)

11. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of Encorafenib, Binimetinib, Ribociclib Metabolite of Binimetinib and Ribociclib: Phase 1b
Time Frame: Phase 1b: Pre dose, 0.5,1.5,2.5,4,6,8 and 24 hr post dose on Day 1 of Cycle 1
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Phase 1b: Encorafenib 50 mg + Binimetinib 45 mg | Phase 1b: Encorafenib 100 mg+ Binimetinib 45 mg | Phase 1b: Encorafenib 200 mg + Binimetinib 45 mg | Phase 1b: Encorafenib 400 mg+ Binimetinib 45 mg | Phase 1b: Encorafenib 450 mg+ Binimetinib 45 mg | Phase 1b: Encorafenib 600 mg+ Binimetinib 45 mg | Phase 1b: Encorafenib 800 mg + Binimetinib 45 mg | Phase 1b: Encorafenib 200 mg+ Binimetinib 45 mg+ Ribociclib 100 mg | Phase 1b: Encorafenib 200 mg+ Binimetinib 45 mg+ Ribociclib 200 mg | Phase 1b: Encorafenib 200 mg+ Binimetinib 45 mg+ Ribociclib 400 mg | Phase 1b: Encorafenib 200 mg+ Binimetinib 45 mg+ Ribociclib 600 mg
Number analyzed (Participants) | 6 | 5 | 4 | 5 | 13 | 8 | 6 | 4 | 5 | 6 | 6
ng/mL
  Encorafenib: number analyzed (Participants) | 6 | 5 | 4 | 4 | 13 | 7 | 6 | 4 | 5 | 6 | 6
  Encorafenib | 855 (480) | 1930 (652) | 3820 (1550) | 6930 (1950) | 7620 (3350) | 10300 (3170) | 7880 (2910) | 2920 (499) | 3190 (1010) | 3450 (1140) | 4200 (1020)
  Binimetinib: number analyzed (Participants) | 6 | 5 | 3 | 4 | 13 | 7 | 4 | 4 | 5 | 6 | 6
  Binimetinib | 635 (402) | 587 (147) | 986 (771) | 532 (227) | 807 (398) | 901 (480) | 621 (160) | 462 (85.6) | 867 (232) | 560 (213) | 703 (222)
  Ribociclib: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 5 | 6 | 6
  Ribociclib |  |  |  |  |  |  |  | 74.2 (37.5) | 219 (95.2) | 554 (251) | 1220 (701)
  Metabolite of Binimetinib: number analyzed (Participants) | 6 | 5 | 3 | 4 | 13 | 7 | 4 | 4 | 5 | 6 | 6
  Metabolite of Binimetinib | 79.3 (55.3) | 75.3 (10.7) | 90.8 (88.0) | 67.9 (32.0) | 85.1 (34.9) | 93.5 (67.0) | 81.1 (32.4) | 41.8 (13.2) | 83.2 (28.2) | 40.2 (22.3) | 45.0 (25.4)
  Metabolite of Ribociclib: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 5 | 6 | 6
  Metabolite of Ribociclib |  |  |  |  |  |  |  | 5.90 (1.73) | 28.7 (7.82) | 58.0 (39.6) | 73.8 (24.3)

12. Secondary Outcome: Cmax at Steady State (Cmax,ss) of Encorafenib, Binimetinib, Ribociclib, Metabolite of Binimetinib and Ribociclib: Phase 1b
Time Frame: Phase 1b: Pre dose,0.5,1.5,2.5,4,6,8 and 24 hr post dose on Day 15 of Cycle 1
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Phase 1b: Encorafenib 50 mg+ Binimetinib 45 mg | Phase 1b: Encorafenib 100 mg + Binimetinib 45 mg | Phase 1b: Encorafenib 200 mg+ Binimetinib 45 mg | Phase 1b: Encorafenib 400 mg+ Binimetinib 45 mg | Phase 1b: Encorafenib 450 mg+ Binimetinib 45 mg | Phase 1b: Encorafenib 600 mg+ Binimetinib 45 mg | Phase 1b: Encorafenib 800 mg+ Binimetinib 45 mg | Phase 1b: Encorafenib 200 mg+ Binimetinib 45 mg+ Ribociclib 100 mg | Phase 1b: Encorafenib 200 mg+ Binimetinib 45 mg+ Ribociclib 200 mg | Phase 1b: Encorafenib 200 mg+ Binimetinib 45 mg+ Ribociclib 400 mg | Phase 1b: Encorafenib 200 mg+ Binimetinib 45 mg+ Ribociclib 600 mg
Number analyzed (Participants) | 6 | 5 | 4 | 5 | 13 | 8 | 6 | 4 | 5 | 6 | 6
ng/mL
  Encorafenib: number analyzed (Participants) | 6 | 5 | 2 | 3 | 11 | 6 | 6 | 4 | 5 | 5 | 5
  Encorafenib | 587 (321) | 1190 (409) | 1060 (194) | 3760 (1380) | 4320 (2260) | 11100 (14100) | 7320 (2700) | 1670 (453) | 2320 (779) | 2480 (1090) | 2590 (929)
  Binimetinib: number analyzed (Participants) | 6 | 5 | 2 | 4 | 11 | 6 | 5 | 4 | 4 | 5 | 5
  Binimetinib | 693 (283) | 568 (233) | 616 (438) | 553 (336) | 638 (283) | 716 (321) | 726 (206) | 584 (181) | 778 (160) | 563 (262) | 609 (261)
  Ribociclib: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 5 | 5 | 5
  Ribociclib |  |  |  |  |  |  |  | 43.7 (16.1) | 146 (111) | 493 (258) | 752 (304)
  Metabolite of Binimetinib: number analyzed (Participants) | 6 | 5 | 2 | 4 | 11 | 6 | 5 | 4 | 4 | 5 | 5
  Metabolite of Binimetinib | 39.7 (43.7) | 36.0 (25.9) | 27.3 (12.6) | 31.7 (25.9) | 38.8 (21.8) | 35.0 (25.3) | 47.3 (19.5) | 38.3 (25.4) | 55.1 (26.5) | 33.2 (16.7) | 33.7 (12.8)
  Metabolite of Ribociclib: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 5 | 5 | 5
  Metabolite of Ribociclib |  |  |  |  |  |  |  | 16.8 (9.77) | 49.7 (19.5) | 155 (30.5) | 195 (56.3)

13. Secondary Outcome: Elimination Half-life (t1/2) of Encorafenib, Binimetinib, Ribociclib, Metabolite of Binimetinib and Ribociclib: Phase 1b
Time Frame: Phase 1b: Pre dose, 0.5,1.5,2.5,4,6,8 and 24 hr post dose on Day 1 of Cycle 1
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Hour
Arm/Group | Phase 1b: Encorafenib 50 mg+ Binimetinib 45 mg | Phase 1b: Encorafenib 100 mg+ Binimetinib 45 mg | Phase 1b: Encorafenib 200 mg + Binimetinib 45 mg | Phase 1b: Encorafenib 400 mg+ Binimetinib 45 mg | Phase 1b: Encorafenib 450 mg + Binimetinib 45 mg | Phase 1b: Encorafenib 600 mg + Binimetinib 45 mg | Phase 1b: Encorafenib 800 mg+ Binimetinib 45 mg | Phase 1b: Encorafenib 200 mg+ Binimetinib 45 mg+ Ribociclib 100 mg | Phase 1b: Encorafenib 200 mg+ Binimetinib 45 mg+ Ribociclib 200 mg | Phase 1b: Encorafenib 200 mg+ Binimetinib 45 mg+ Ribociclib 400 mg | Phase 1b: Encorafenib 200 mg+ Binimetinib 45 mg+ Ribociclib 600 mg
Number analyzed (Participants) | 6 | 5 | 4 | 5 | 13 | 8 | 6 | 4 | 5 | 6 | 6
Hour
  Encorafenib: number analyzed (Participants) | 6 | 5 | 4 | 4 | 13 | 7 | 5 | 4 | 4 | 3 | 5
  Encorafenib | 3.68 (0.605) | 3.65 (0.351) | 2.88 (0.121) | 4.19 (2.13) | 3.47 (0.402) | 3.21 (0.550) | 3.04 (0.0935) | 3.25 (0.375) | 2.10 (0.451) | 2.95 (1.13) | 2.59 (0.567)
  Binimetinib: number analyzed (Participants) | 5 | 4 | 3 | 3 | 11 | 7 | 4 | 4 | 4 | 3 | 4
  Binimetinib | 2.36 (0.427) | 2.37 (0.704) | 2.10 (0.522) | 2.51 (0.472) | 2.22 (0.439) | 2.12 (0.314) | 1.99 (0.601) | 3.73 (1.78) | 2.45 (1.19) | 3.11 (1.01) | 1.98 (0.523)
  Ribociclib: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 5 | 4 | 4
  Ribociclib |  |  |  |  |  |  |  | 8.71 (2.32) | 7.97 (1.24) | 10.3 (3.94) | 7.71 (0.408)
  Metabolite of Binimetinib: number analyzed (Participants) | 5 | 3 | 2 | 3 | 9 | 5 | 4 | 3 | 4 | 0 | 4
  Metabolite of Binimetinib | 2.82 (0.757) | 2.00 (0.0542) | 2.95 (0.739) | 2.58 (0.737) | 2.64 (0.604) | 2.28 (0.546) | 2.37 (0.517) | 3.39 (1.57) | 2.49 (0.528) |  | 2.32 (0.455)
  Metabolite of Ribociclib: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 1 | 1
  Metabolite of Ribociclib |  |  |  |  |  |  |  | 23.2 (NA) — Standard deviation could not be calculated as only 1 participant was evaluable. | 15.4 (6.92) | 7.99 (NA) — Standard deviation could not be calculated as only 1 participant was evaluable. | 15.9 (NA) — Standard deviation could not be calculated as only 1 participant was evaluable.

14. Secondary Outcome: t1/2 at Steady State (t1/2,ss) of Encorafenib, Binimetinib, Ribociclib, Metabolite of Binimetinib and Ribociclib: Phase 1b
Time Frame: Phase 1b: Pre dose,0.5,1.5,2.5,4,6,8 and 24 hr post dose on Day 15 of Cycle 1
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Hour
Arm/Group | Phase 1b: Encorafenib 50 mg + Binimetinib 45 mg | Phase 1b: Encorafenib 100 mg+ Binimetinib 45 mg | Phase 1b: Encorafenib 200 mg+ Binimetinib 45 mg | Phase 1b: Encorafenib 400 mg + Binimetinib 45 mg | Phase 1b: Encorafenib 450 mg + Binimetinib 45 mg | Phase 1b: Encorafenib 600 mg + Binimetinib 45 mg | Phase 1b: Encorafenib 800 mg+ Binimetinib 45 mg | Phase 1b: Encorafenib 200 mg+ Binimetinib 45 mg+ Ribociclib 100 mg | Phase 1b: Encorafenib 200 mg+ Binimetinib 45 mg+ Ribociclib 200 mg | Phase 1b: Encorafenib 200 mg+ Binimetinib 45 mg+ Ribociclib 400 mg | Phase 1b: Encorafenib 200 mg+ Binimetinib 45 mg+ Ribociclib 600 mg
Number analyzed (Participants) | 6 | 5 | 4 | 5 | 13 | 8 | 6 | 4 | 5 | 6 | 6
Hour
  Encorafenib: number analyzed (Participants) | 5 | 4 | 2 | 3 | 11 | 6 | 6 | 4 | 5 | 5 | 4
  Encorafenib | 4.74 (1.18) | 4.47 (0.380) | 4.32 (1.25) | 4.21 (0.724) | 3.57 (0.688) | 3.40 (0.223) | 3.37 (0.511) | 3.98 (0.331) | 3.24 (0.776) | 4.00 (0.922) | 3.52 (0.237)
  Binimetinib: number analyzed (Participants) | 2 | 4 | 1 | 4 | 9 | 0 | 3 | 3 | 3 | 4 | 4
  Binimetinib | 4.74 (1.43) | 4.80 (1.40) | 3.28 (NA) — Standard deviation could not be calculated as only 1 participant was evaluable. | 4.20 (1.36) | 3.61 (1.14) |  | 2.91 (0.157) | 4.04 (2.03) | 2.67 (1.40) | 3.69 (1.16) | 5.21 (1.75)
  Ribociclib: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 4 | 4 | 3
  Ribociclib |  |  |  |  |  |  |  | 13.2 (2.26) | 11.4 (6.07) | 8.49 (2.80) | 10.3 (5.32)
  Metabolite of Binimetinib: number analyzed (Participants) | 2 | 2 | 1 | 1 | 5 | 2 | 3 | 1 | 3 | 2 | 2
  Metabolite of Binimetinib | 4.51 (1.23) | 7.23 (5.44) | 2.07 (NA) — Standard deviation could not be calculated as only 1 participant was evaluable. | 4.61 (NA) — Standard deviation could not be calculated as only 1 participant was evaluable. | 2.79 (1.23) | 4.06 (0.195) | 3.33 (0.524) | 5.12 (NA) — Standard deviation could not be calculated as only 1 participant was evaluable. | 2.58 (0.626) | 3.44 (0.115) | 4.38 (2.14)
  Metabolite of Ribociclib: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 4 | 2 | 2
  Metabolite of Ribociclib |  |  |  |  |  |  |  | 18.3 (3.23) | 15.7 (6.62) | 15.0 (6.27) | 18.6 (2.76)

15. Secondary Outcome: Accumulation Ratio (RA) of Encorafenib, Binimetinib, Ribociclib Metabolite of Binimetinib and Ribociclib: Phase 1b
Description: Accumulation ratio was calculated as AUCtau,ss/AUCtau.
Time Frame: Phase 1b: Pre dose, 0.5,1.5,2.5,4,6,8 and 24 hr post dose on Day 1 and 15 of Cycle 1
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Phase 1b: Encorafenib 50 mg+ Binimetinib 45 mg | Phase 1b: Encorafenib 100 mg+ Binimetinib 45 mg | Phase 1b: Encorafenib 200 mg+ Binimetinib 45 mg | Phase 1b: Encorafenib 400 mg+ Binimetinib 45 mg | Phase 1b: Encorafenib 450 mg + Binimetinib 45 mg | Phase 1b: Encorafenib 600 mg+ Binimetinib 45 mg | Phase 1b: Encorafenib 800 mg+ Binimetinib 45 mg | Phase 1b: Encorafenib 200 mg+ Binimetinib 45 mg+ Ribociclib 100 mg | Phase 1b: Encorafenib 200 mg+ Binimetinib 45 mg+ Ribociclib 200 mg | Phase 1b: Encorafenib 200 mg+ Binimetinib 45 mg+ Ribociclib 400 mg | Phase 1b: Encorafenib 200 mg+ Binimetinib 45 mg+ Ribociclib 600 mg
Number analyzed (Participants) | 6 | 5 | 4 | 5 | 13 | 8 | 6 | 4 | 5 | 6 | 6
Ratio
  Encorafenib: number analyzed (Participants) | 6 | 5 | 2 | 3 | 11 | 6 | 5 | 4 | 4 | 3 | 4
  Encorafenib | 0.857 (0.351) | 0.601 (0.322) | 0.298 (0.0682) | 0.348 (0.125) | 0.458 (0.188) | 0.473 (0.215) | 0.690 (0.291) | 0.460 (0.134) | 0.841 (0.178) | 0.833 (0.463) | 0.806 (0.393)
  Binimetinib: number analyzed (Participants) | 5 | 4 | 2 | 4 | 9 | 6 | 4 | 4 | 3 | 2 | 4
  Binimetinib | 1.51 (0.248) | 1.26 (0.152) | 1.07 (0.142) | 0.989 (0.353) | 1.03 (0.339) | 0.969 (0.297) | 1.19 (0.472) | 1.29 (0.572) | 0.778 (0.102) | 1.19 (0.324) | 1.08 (0.316)
  Ribociclib: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 5 | 5 | 5
  Ribociclib |  |  |  |  |  |  |  | 0.640 (0.282) | 0.734 (0.404) | 1.11 (0.753) | 0.712 (0.168)
  Metabolite of Binimetinib: number analyzed (Participants) | 3 | 1 | 1 | 2 | 4 | 1 | 3 | 1 | 3 | 0 | 4
  Metabolite of Binimetinib | 0.899 (0.542) | 0.588 (NA) — Standard deviation could not be calculated as only 1 participant was evaluable. | 0.285 (NA) — Standard deviation could not be calculated as only 1 participant was evaluable. | 0.954 (0.0302) | 0.546 (0.300) | 0.499 (NA) — Standard deviation could not be calculated as only 1 participant was evaluable. | 0.569 (0.0381) | 1.56 (NA) — Standard deviation could not be calculated as only 1 participant was evaluable. | 0.726 (0.194) |  | 0.910 (0.195)
  Metabolite of Ribociclib: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 5 | 5 | 5
  Metabolite of Ribociclib |  |  |  |  |  |  |  | 2.81 (0.619) | 1.93 (0.684) | 2.73 (0.517) | 2.97 (0.548)

16. Secondary Outcome: Objective Response Rate (ORR): Phase 1b
Description: ORR was defined as the percentage of participants with a best overall response of CR or PR. As per RECIST v1.1, CR was defined as complete disappearance of all target lesions and non-target disease. All nodes, both target and non-target, must have a reduction in short axis <10 mm. PR was defined as >= 30 % decrease under baseline of sum of diameters of all target lesions taking as reference the baseline sum of diameters.
Time Frame: Phase 1b: From Day 1 of dosing till complete response or partial response achieved (maximum exposure of treatment in Phase 1b was 118.3 months)
Population: FAS included all participants who received at least one dose of LGX818 or MEK162 or LEE011.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Phase 1b: Encorafenib 50 mg+ Binimetinib 45 mg | Phase 1b: Encorafenib 100 mg+ Binimetinib 45 mg | Phase 1b: Encorafenib 200 mg+ Binimetinib 45 mg | Phase 1b: Encorafenib 400 mg+ Binimetinib 45 mg | Phase 1b: Encorafenib 450 mg+ Binimetinib 45 mg | Phase 1b: Encorafenib 600 mg+ Binimetinib 45 mg | Phase 1b: Encorafenib 800 mg+ Binimetinib 45 mg | Phase 1b: Encorafenib 200 mg+ Binimetinib 45 mg+ Ribociclib 100 mg | Phase 1b: Encorafenib 200 mg+ Binimetinib 45 mg+ Ribociclib 200 mg | Phase 1b: Encorafenib 200 mg+ Binimetinib 45 mg+ Ribociclib 400 mg | Phase 1b: Encorafenib 200 mg+ Binimetinib 45 mg+ Ribociclib 600 mg
Number analyzed (Participants) | 6 | 5 | 4 | 5 | 13 | 8 | 6 | 4 | 5 | 6 | 6
Percentage of participants | 66.7 [22.3 to 95.7] | 40.0 [5.3 to 85.3] | 25.0 [0.6 to 80.6] | 40.0 [5.3 to 85.3] | 53.8 [25.1 to 80.8] | 25.0 [3.2 to 65.1] | 50.0 [11.8 to 88.2] | 75.0 [19.4 to 99.4] | 60.0 [14.7 to 94.7] | 66.7 [22.3 to 95.7] | 66.7 [22.3 to 95.7]

17. Secondary Outcome: Progression Free Survival (PFS): Phase 2
Description: PFS was defined as the time from the start of study treatment to the date of the event defined as the first documented progression or death due to any cause. If a participant did not have an event, PFS was censored at the date of last adequate tumor assessment. Per RECIST 1.1, PD= At least a 20% increase in the sum of diameter of all measured target lesions, taking as reference the smallest sum of diameter of all target lesions recorded at or after baseline. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm^2. Unequivocal progression of existing non-target lesions. Kaplan-Meier method was used for analysis.
Time Frame: Phase 2: From start of study drug until documented PD or death due to any cause or censoring date (maximum exposure of treatment in Phase 2 was 111.5 months)
Population: FAS included all participants who received at least one dose of LGX818 or MEK162 or LEE011.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase 2: Arm 1 (mCRC): Encorafenib + Binimetinib | Phase 2: Arm 2 (Prior BRAFi Melanoma): Encorafenib + Binimetinib | Phase 2: Arm 3 (BRAFi-naïve Melanoma): Encorafenib + Binimetinib | Phase 2: Arm A (BRAFi-naïve Melanoma): Encorafenib + Binimetinib + Ribociclib
Number analyzed (Participants) | 11 | 26 | 42 | 42
Months | 5.4 [2.1 to 9.0] | 3.8 [3.4 to 9.3] | 7.5 [5.7 to 12.2] | 9.0 [5.6 to 11.1]

18. Secondary Outcome: Time to Response (TTR): Phase 2
Description: TTR was defined as the time from the first dose of study treatment to the first documentation of objective tumor response documented in participants with confirmed objective response (CR or PR). As per RECIST v1.1, CR was defined as complete disappearance of all target lesions and non-target disease. All nodes, both target and non-target, must have a reduction in short axis <10 mm. PR was defined as >= 30 % decrease under baseline of sum of diameters of all target lesions taking as reference the baseline sum of diameters. Kaplan-Meier method was used for analysis.
Time Frame: Phase 2: From date of start of treatment until date of first documentation of objective tumor response (maximum exposure of treatment in Phase 2 was 111.5 months)
Population: FAS evaluated.Here "Number of Participants Analyzed" signifies the number of participants who were confirmed responders and were evaluable for this outcome measure.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase 2: Arm 1 (mCRC): Encorafenib + Binimetinib | Phase 2: Arm 2 (Prior BRAFi Melanoma): Encorafenib + Binimetinib | Phase 2: Arm 3 (BRAFi-naïve Melanoma): Encorafenib + Binimetinib | Phase 2: Arm A (BRAFi-naïve Melanoma): Encorafenib + Binimetinib + Ribociclib
Number analyzed (Participants) | 2 | 11 | 28 | 25
Months | 2.6 [1.6 to 3.6] | 1.8 [1.0 to 5.6] | 1.0 [1.0 to 1.8] | 1.9 [1.8 to 2.1]

19. Secondary Outcome: Duration of Response (DOR): Phase 2
Description: DOR was defined as the time from the first documentation of objective tumor response to the first documentation of objective tumor progression or to death due to underlying cancer, whichever occurred first in participants with confirmed objective response (CR or PR). As per RECIST v1.1, CR was defined as complete disappearance of all target lesions and non-target disease. All nodes, both target and non-target, must have a reduction in short axis <10 mm. PR was defined as >= 30 % decrease under baseline of sum of diameters of all target lesions taking as reference the baseline sum of diameters. Kaplan-Meier method was used for analysis.
Time Frame: Phase 2: From date of first documentation of objective tumor response to the first documentation of objective tumor progression or to death due to underlying cancer, whichever occurred first (maximum exposure of treatment in Phase 2 was 111.5 months)
Population: as for outcome 18
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase 2: Arm 1 (mCRC): Encorafenib + Binimetinib | Phase 2: Arm 2 (Prior BRAFi Melanoma): Encorafenib + Binimetinib | Phase 2: Arm 3 (BRAFi-naïve Melanoma): Encorafenib + Binimetinib | Phase 2: Arm A (BRAFi-naïve Melanoma): Encorafenib + Binimetinib + Ribociclib
Number analyzed (Participants) | 2 | 11 | 28 | 25
Months | 7.1 [3.8 to NA] — Upper limit of CI could not be estimated because of insufficient number of participants with this event and hence could not be reported. | 3.8 [2.9 to 12.9] | 10.9 [6.5 to 19.5] | 7.5 [5.6 to 25.8]

20. Secondary Outcome: Overall Survival (OS): Phase 2
Description: OS was defined as the time from date of randomization/start of treatment to date of death due to any cause. If a participant was not known to have died, survival was censored at the date of last contact. Analysis was performed using Kaplan-Meier method.
Time Frame: Phase 2: From date of start of study treatment until date of death or censoring date (maximum exposure of treatment in Phase 2 was 111.5 months)
Population: FAS included all participants who received at least one dose of LGX818 or MEK162 or LEE011.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase 2: Arm 1 (mCRC): Encorafenib + Binimetinib | Phase 2: Arm 2 (Prior BRAFi Melanoma): Encorafenib + Binimetinib | Phase 2: Arm 3 (BRAFi-naïve Melanoma): Encorafenib + Binimetinib | Phase 2: Arm A (BRAFi-naïve Melanoma): Encorafenib + Binimetinib + Ribociclib
Number analyzed (Participants) | 11 | 26 | 42 | 42
Months | 9.5 [7.7 to 27.2] | 11.4 [5.9 to 20.7] | 23.1 [17.3 to NA] — Upper limit of CI could not be estimated because of insufficient number of participants with this event and hence could not be reported. | 21.8 [14.8 to 35.7]

21. Secondary Outcome: Number of Participants With Molecular Alterations of Tumor Tissues Using Potential Predictive Markers: Phase 1b
Description: Molecular alterations of tumor tissues was determined using the following potential predictive markers: Biomarkers like V-raf murine sarcoma viral oncogene homolog B1 (BRAF),V-Ki-ras2 Kirsten rat sarcoma viral oncogene homolog (KRAS), Phosphatase and tensin homolog (PTEN), Phosphatidylinositol 3' kinase catalytic alphapolypeptide (PIK3CA), Epidermal growth factor receptor (EGFR).
Time Frame: Phase 1b: Baseline
Population: FAS included all participants who received at least one dose of LGX818 or MEK162 or LEE011.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1b: Encorafenib 50 mg+ Binimetinib 45 mg | Phase 1b: Encorafenib 100 mg+ Binimetinib 45 mg | Phase 1b: Encorafenib 200 mg+ Binimetinib 45 mg | Phase 1b: Encorafenib 400 mg+ Binimetinib 45 mg | Phase 1b: Encorafenib 450 mg+ Binimetinib 45 mg | Phase 1b: Encorafenib 600 mg+ Binimetinib 45 mg | Phase 1b: Encorafenib 800 mg+ Binimetinib 45 mg | Phase 1b: Encorafenib 200 mg + Binimetinib 45 mg+ Ribociclib 100 mg | Phase 1b: Encorafenib 200 mg + Binimetinib 45 mg+ Ribociclib 200 mg | Phase 1b: Encorafenib 200 mg + Binimetinib 45 mg+ Ribociclib 400 mg | Phase 1b: Encorafenib 200 mg + Binimetinib 45 mg+ Ribociclib 600 mg
Number analyzed (Participants) | 6 | 5 | 4 | 5 | 13 | 8 | 6 | 4 | 5 | 6 | 6
Participants
  BRAF | 5 | 4 | 3 | 4 | 7 | 7 | 3 | 3 | 4 | 5 | 4
  KRAS | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  PTEN | 0 | 1 | 0 | 0 | 1 | 2 | 1 | 0 | 0 | 0 | 1
  PIK3CA | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  EGFR | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0

22. Secondary Outcome: Number of Participants With Molecular Alterations of Tumor Tissues Using Potential Predictive Markers: Phase 2
Description: Molecular alterations of tumor tissues was determined using the following potential predictive markers: BRAF, HRAS, KRAS, Neuroblastoma RAS viral oncogene homolog (NRAS), PTEN, PIK3CA, Mitogen-activated protein kinase 1 (MAP2K1), Mitogen-activated protein kinase 2 (MAP2K2), EGFR.
Time Frame: Phase 2: Baseline
Population: FAS included all participants who received at least one dose of LGX818 or MEK162 or LEE011.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2: Arm 1 (mCRC): Encorafenib + Binimetinib | Phase 2: Arm 2 (Prior BRAFi Melanoma): Encorafenib + Binimetinib | Phase 2: Arm 3 (BRAFi-naïve Melanoma): Encorafenib + Binimetinib | Phase 2: Arm A (BRAFi-naïve Melanoma): Encorafenib + Binimetinib + Ribociclib
Number analyzed (Participants) | 11 | 26 | 42 | 42
Participants
  BRAF | 4 | 15 | 20 | 30
  HRAS | 0 | 0 | 0 | 0
  KRAS | 2 | 0 | 0 | 0
  NRAS | 0 | 2 | 0 | 0
  PTEN | 1 | 6 | 5 | 5
  PIK3CA | 2 | 0 | 0 | 2
  MAP2K1 | 0 | 3 | 1 | 0
  MAP2K2 | 0 | 0 | 0 | 0
  ARAF | 0 | 0 | 0 | 0
  EGFR | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Day 1 of dosing up to 30 days after last dose (maximum treatment exposure for Phase 1b was 118.3 months, Phase 2 was 111.5 months)
Description: Same event may appear as both non-SAE and SAE, but what is presented are distinct events. An event may be categorized as serious in 1 participant and non-serious in other participant, or a participant may have experienced both SAE and non-SAE. Safety analysis set was evaluated.
Arm/Group | Phase 1b: Encorafenib 50 mg + Binimetinib 45 mg | Phase 1b: Encorafenib 100 mg+ Binimetinib 45 mg | Phase 1b: Encorafenib 200 mg + Binimetinib 45 mg | Phase 1b: Encorafenib 400 mg + Binimetinib 45 mg | Phase 1b: Encorafenib 450 mg+ Binimetinib 45 mg | Phase 1b: Encorafenib 600 mg + Binimetinib 45 mg | Phase 1b: Encorafenib 800 mg + Binimetinib 45 mg | Phase 1b: Encorafenib 200 mg+ Binimetinib 45 mg+ Ribociclib 100 mg | Phase 1b: Encorafenib 200 mg+ Binimetinib 45 mg+ Ribociclib 200 mg | Phase 1b: Encorafenib 200 mg+ Binimetinib 45 mg+ Ribociclib 400 mg | Phase 1b: Encorafenib 200 mg+ Binimetinib 45 mg + Ribociclib 600 mg | Phase 2: Arm 1 (mCRC): Encorafenib + Binimetinib | Phase 2: Arm 2 (Prior BRAFi Melanoma): Encorafenib + Binimetinib | Phase 2: Arm 3 (BRAFi-naïve Melanoma): Encorafenib + Binimetinib | Phase 2: Arm A (BRAFi-naïve Melanoma): Encorafenib + Binimetinib + Ribociclib
All-Cause Mortality (participants affected / at risk) | 1/6 | 0/5 | 1/4 | 2/5 | 2/13 | 0/8 | 1/6 | 0/4 | 1/5 | 0/6 | 2/6 | 9/11 | 22/26 | 22/42 | 28/42
Serious Adverse Events (participants affected / at risk) | 4/6 | 2/5 | 2/4 | 2/5 | 5/13 | 4/8 | 4/6 | 2/4 | 3/5 | 3/6 | 2/6 | 5/11 | 13/26 | 18/42 | 21/42
Other Adverse Events (participants affected / at risk) | 6/6 | 5/5 | 4/4 | 5/5 | 13/13 | 8/8 | 6/6 | 4/4 | 5/5 | 5/6 | 6/6 | 11/11 | 26/26 | 39/42 | 42/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1b: Encorafenib 50 mg + Binimetinib 45 mg (N=6) | Phase 1b: Encorafenib 100 mg+ Binimetinib 45 mg (N=5) | Phase 1b: Encorafenib 200 mg + Binimetinib 45 mg (N=4) | Phase 1b: Encorafenib 400 mg + Binimetinib 45 mg (N=5) | Phase 1b: Encorafenib 450 mg+ Binimetinib 45 mg (N=13) | Phase 1b: Encorafenib 600 mg + Binimetinib 45 mg (N=8) | Phase 1b: Encorafenib 800 mg + Binimetinib 45 mg (N=6) | Phase 1b: Encorafenib 200 mg+ Binimetinib 45 mg+ Ribociclib 100 mg (N=4) | Phase 1b: Encorafenib 200 mg+ Binimetinib 45 mg+ Ribociclib 200 mg (N=5) | Phase 1b: Encorafenib 200 mg+ Binimetinib 45 mg+ Ribociclib 400 mg (N=6) | Phase 1b: Encorafenib 200 mg+ Binimetinib 45 mg + Ribociclib 600 mg (N=6) | Phase 2: Arm 1 (mCRC): Encorafenib + Binimetinib (N=11) | Phase 2: Arm 2 (Prior BRAFi Melanoma): Encorafenib + Binimetinib (N=26) | Phase 2: Arm 3 (BRAFi-naïve Melanoma): Encorafenib + Binimetinib (N=42) | Phase 2: Arm A (BRAFi-naïve Melanoma): Encorafenib + Binimetinib + Ribociclib (N=42)
Intracardiac mass (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vertigo positional (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Retinal detachment (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Retinal vein occlusion (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Retinopathy hypertensive (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 2 | 0 | 0 | 0
Melaena (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 3 | 2 | 2
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 2 | 3
Pyrexia (General disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 3 | 2
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pharyngeal abscess (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Post procedural infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyelonephritis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Septic shock (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Streptococcal bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pubis fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Traumatic haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bone disorder (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chronic myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Balance disorder (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cerebral infarction (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemorrhage intracranial (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hemiparesis (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nerve root compression (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Seizure (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Suicide attempt (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pericarditis (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Blindness (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Eye pain (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Iritis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Visual impairment (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Detachment of retinal pigment epithelium (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Macular oedema (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 1
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gastrointestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Axillary pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Chills (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
General physical health deterioration (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2
Disease progression (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hepatic haemorrhage (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Erysipelas (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lung infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Abdominal abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dermo-hypodermitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Polyarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Intracranial tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1
Ataxia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Loss of consciousness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Polyneuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Tremor (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lymphadenectomy (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Aortic stenosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Epilepsy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Troponin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypercreatininaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Mediastinoscopy (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1b: Encorafenib 50 mg + Binimetinib 45 mg (N=6) | Phase 1b: Encorafenib 100 mg+ Binimetinib 45 mg (N=5) | Phase 1b: Encorafenib 200 mg + Binimetinib 45 mg (N=4) | Phase 1b: Encorafenib 400 mg + Binimetinib 45 mg (N=5) | Phase 1b: Encorafenib 450 mg+ Binimetinib 45 mg (N=13) | Phase 1b: Encorafenib 600 mg + Binimetinib 45 mg (N=8) | Phase 1b: Encorafenib 800 mg + Binimetinib 45 mg (N=6) | Phase 1b: Encorafenib 200 mg+ Binimetinib 45 mg+ Ribociclib 100 mg (N=4) | Phase 1b: Encorafenib 200 mg+ Binimetinib 45 mg+ Ribociclib 200 mg (N=5) | Phase 1b: Encorafenib 200 mg+ Binimetinib 45 mg+ Ribociclib 400 mg (N=6) | Phase 1b: Encorafenib 200 mg+ Binimetinib 45 mg + Ribociclib 600 mg (N=6) | Phase 2: Arm 1 (mCRC): Encorafenib + Binimetinib (N=11) | Phase 2: Arm 2 (Prior BRAFi Melanoma): Encorafenib + Binimetinib (N=26) | Phase 2: Arm 3 (BRAFi-naïve Melanoma): Encorafenib + Binimetinib (N=42) | Phase 2: Arm A (BRAFi-naïve Melanoma): Encorafenib + Binimetinib + Ribociclib (N=42)
Anaemia (Blood and lymphatic system disorders) | 1 | 1 | 1 | 1 | 1 | 3 | 0 | 1 | 1 | 2 | 2 | 1 | 6 | 7 | 11
Neutropenia (Blood and lymphatic system disorders) | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 2 | 0 | 0 | 0 | 17
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 3
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 3
Detachment of retinal pigment epithelium (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 2 | 1 | 2 | 0 | 7 | 5 | 2
Macular oedema (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 2 | 2 | 1 | 1 | 4 | 3 | 5
Retinal detachment (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 5
Chorioretinopathy (Eye disorders) | 1 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 3 | 2 | 0
Photophobia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 3 | 0
Retinopathy (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 7 | 4 | 6 | 9
Subretinal fluid (Eye disorders) | 0 | 0 | 0 | 1 | 4 | 1 | 1 | 1 | 2 | 2 | 1 | 0 | 4 | 9 | 3
Vision blurred (Eye disorders) | 3 | 1 | 1 | 1 | 1 | 2 | 3 | 0 | 0 | 0 | 0 | 1 | 5 | 12 | 0
Visual impairment (Eye disorders) | 1 | 0 | 0 | 2 | 1 | 2 | 1 | 2 | 1 | 0 | 1 | 0 | 4 | 3 | 6
Cataract (Eye disorders) | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dry eye (Eye disorders) | 1 | 0 | 1 | 0 | 3 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 3 | 2 | 0 | 2 | 4 | 2 | 3 | 1 | 0 | 2 | 2 | 0 | 2 | 11 | 6
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 1 | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5
Constipation (Gastrointestinal disorders) | 3 | 3 | 2 | 2 | 4 | 3 | 4 | 2 | 0 | 1 | 1 | 4 | 5 | 13 | 12
Diarrhoea (Gastrointestinal disorders) | 4 | 1 | 1 | 2 | 7 | 7 | 4 | 0 | 1 | 3 | 4 | 8 | 14 | 20 | 18
Dry mouth (Gastrointestinal disorders) | 2 | 2 | 0 | 0 | 3 | 0 | 1 | 0 | 2 | 1 | 1 | 0 | 1 | 4 | 4
Dyspepsia (Gastrointestinal disorders) | 0 | 2 | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 7 | 2
Nausea (Gastrointestinal disorders) | 3 | 4 | 2 | 2 | 7 | 5 | 3 | 2 | 2 | 0 | 2 | 6 | 11 | 20 | 17
Vomiting (Gastrointestinal disorders) | 2 | 1 | 4 | 2 | 7 | 3 | 1 | 0 | 2 | 0 | 2 | 7 | 9 | 14 | 16
Abdominal distension (Gastrointestinal disorders) | 1 | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 0
Flatulence (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0
Retinal degeneration (Eye disorders) | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Retinal haemorrhage (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vitreous detachment (Eye disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vitreous floaters (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Asthenia (General disorders) | 0 | 1 | 0 | 1 | 1 | 1 | 1 | 0 | 2 | 1 | 2 | 7 | 3 | 3 | 9
Fatigue (General disorders) | 4 | 2 | 0 | 2 | 7 | 3 | 3 | 2 | 1 | 1 | 2 | 2 | 10 | 12 | 14
Influenza like illness (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 4 | 3
Oedema peripheral (General disorders) | 2 | 1 | 0 | 0 | 1 | 2 | 1 | 1 | 0 | 1 | 2 | 0 | 4 | 7 | 3
Chills (General disorders) | 1 | 0 | 0 | 1 | 3 | 1 | 1 | 0 | 0 | 1 | 0 | 2 | 5 | 7 | 4
Pyrexia (General disorders) | 4 | 0 | 1 | 1 | 4 | 1 | 0 | 2 | 3 | 1 | 1 | 6 | 4 | 14 | 12
Peripheral swelling (General disorders) | 1 | 1 | 1 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 0
Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4
Oral herpes (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Upper respiratory tract infection (Infections and infestations) | 2 | 1 | 0 | 1 | 2 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 2
Nasopharyngitis (Infections and infestations) | 2 | 2 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 4 | 4 | 2 | 0
Influenza (Infections and infestations) | 2 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0 | 1 | 2 | 2 | 3 | 2 | 1 | 1 | 1 | 1 | 1 | 5 | 11 | 11
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 1 | 2 | 1 | 3 | 1 | 1 | 1 | 2 | 1 | 1 | 6 | 12 | 10
Blood creatine phosphokinase increased (Investigations) | 3 | 2 | 0 | 1 | 0 | 1 | 1 | 1 | 3 | 3 | 2 | 0 | 6 | 15 | 11
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 1 | 7 | 9
Haemoglobin decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 0 | 0 | 0 | 0
Lipase increased (Investigations) | 1 | 0 | 0 | 0 | 3 | 1 | 1 | 0 | 0 | 1 | 0 | 1 | 1 | 14 | 4
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4
Platelet count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 4
White blood cell count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 3 | 4
Amylase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 6 | 0
Ejection fraction decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 0
Weight increased (Investigations) | 1 | 0 | 0 | 1 | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 6 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 6 | 12 | 0
Weight decreased (Investigations) | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 0 | 1 | 3 | 1 | 1 | 0 | 0 | 4 | 1 | 4 | 8
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 4 | 3
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 1 | 3 | 3
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 3 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 6 | 0
Hypercreatininaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 0
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 2 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 1 | 0 | 2 | 0 | 1 | 0 | 0 | 1 | 2 | 2 | 5
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 3 | 4 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 3 | 0
Iron deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 3 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 3 | 0 | 0 | 2 | 1 | 2 | 2 | 3 | 0 | 2 | 4 | 7 | 15 | 6
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 1 | 1 | 2 | 2 | 1 | 0 | 1 | 0 | 1 | 4 | 5 | 8 | 7
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 3 | 2 | 0 | 2 | 0 | 0 | 1 | 1 | 0 | 7 | 4
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 3 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 4 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 2 | 2 | 2 | 3 | 2 | 3 | 0 | 0 | 1 | 2 | 7 | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 1 | 2 | 1 | 2 | 1 | 3 | 2 | 0 | 0 | 1 | 1 | 5 | 5 | 8
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Joint stiffness (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 2 | 0 | 1 | 1 | 2 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 2 | 6
Headache (Nervous system disorders) | 2 | 1 | 1 | 2 | 3 | 2 | 5 | 1 | 1 | 0 | 2 | 1 | 1 | 8 | 10
Dizziness (Nervous system disorders) | 2 | 1 | 0 | 0 | 2 | 2 | 2 | 0 | 0 | 0 | 0 | 2 | 1 | 9 | 0
Paraesthesia (Nervous system disorders) | 2 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 0
Visual field defect (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 3 | 0
Hypoaesthesia (Nervous system disorders) | 1 | 1 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Memory impairment (Nervous system disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Migraine (Nervous system disorders) | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 1 | 1 | 0 | 0 | 0 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 0
Insomnia (Psychiatric disorders) | 1 | 0 | 1 | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 4 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 3 | 0 | 2 | 2 | 1 | 1 | 0 | 1 | 0 | 1 | 3 | 6 | 11 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 1 | 1 | 3 | 1 | 1 | 0 | 0 | 1 | 0 | 1 | 7 | 5
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 2 | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 3 | 0
Pollakiuria (Renal and urinary disorders) | 2 | 0 | 0 | 0 | 3 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 2 | 2 | 0 | 1 | 0 | 2 | 0 | 1 | 1 | 2 | 1 | 1 | 8 | 3
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 1 | 2 | 0 | 3 | 0 | 0 | 0 | 2 | 1 | 4 | 11 | 5
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 5 | 5
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 4
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 2 | 1 | 2 | 0 | 1 | 0 | 2 | 0 | 3 | 12 | 4
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 3 | 1 | 2 | 2 | 1 | 0 | 0 | 0 | 9 | 8 | 7
Hair texture abnormal (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 4 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Palmoplantar keratoderma (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vitiligo (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 3 | 1 | 0 | 0 | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 9 | 9
Flushing (Vascular disorders) | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hot flush (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Disturbance in attention (Nervous system disorders) | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 0
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0 | 0 | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Uveitis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 4
Chest pain (General disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 4 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publication until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2021-03-15): https://cdn.clinicaltrials.gov/large-docs/98/NCT01543698/Prot_000.pdf
  • Statistical Analysis Plan (2023-01-20): https://cdn.clinicaltrials.gov/large-docs/98/NCT01543698/SAP_001.pdf